CLINICAL TRIAL: NCT04181333
Title: TRASTUZUMAB BS for Intravenous Infusion 60 mg [Pfizer], TRASTUZUMAB BS for Intravenous Infusion 150 mg [Pfizer] General Investigation (Unresectable Advanced/Recurrent HER2-Overexpressing Gastric Cancer)
Brief Title: Safety and Efficacy of Trastuzumab BS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3271007
Record Dates: First submitted 2019-11-07; First posted 2019-11-29 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer
Keywords: Recurrent HER2-Overexpressing Gastric Cancer; TRASTUZUMAB BS
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TRASTUZUMAB BS: Unresectable Advanced/Recurrent HER2-Overexpressing Gastric Cancer patients injected TRASTUZUMAB BS
  Interventions: Drug: TRASTUZUMAB BS

INTERVENTIONS:
Drug: TRASTUZUMAB BS — Regimen A or regimen B is used for HER2-overexpressing breast cancer.
  RegimenB is used for HER2-overexpressing unresectable advanced or recurrent gastric cancer in combination with other anti tumor agent(s).
  Regimen A: The recommended dose for trastuzumab (genetical recombination) [Trastuzumab Biosimilar 3] in adult patients is 4 mg/kg (weight) at initial dose and 2 mg/kg after the second dose, in both of them, by IV drip infusion over 90 minutes once daily every week.
  Regimen B: The recommended dose for trastuzumab (genetical recombination) [Trastuzumab Biosimilar 3] in adult patients is 8 mg/kg (weight) at initial dose and 6 mg/kg after the second dose, in both of them, by IV drip infusion over 90 minutes once daily every 3 weeks.
  If the initial dose is well tolerated, the dosing time after the second dose can be shortened up to 30 minutes.

SUMMARY:
To confirm the safety and efficacy of this drug under the actual use

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable advanced/recurrent gastric cancer who are confirmed to have HER2 overexpression and started treatment with this drug*
* Patients who receive this drug* for the first time after this drug* is launched * Not including the biological product, HERCEPTIN, and biosimilars of HERCEPTIN other than this drug

Exclusion Criteria:

- not specified in this study

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 patients
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse drug reactions in this surveillance | 24 weeks

SECONDARY OUTCOMES:
Assessment of tumor response: Assess the tumor response according to RECIST Ver. 1.1. | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3271007